CLINICAL TRIAL: NCT04723953
Title: Cardiac Fibroblast Activation Detected by 68Ga-FAPI PET/MR is a Prognostic Indicator in Patients With Myocardial Infarction.
Brief Title: Cardiac Fibroblast Activation Detected by 68Ga-FAPI PET/MR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: (2020)CER(152)
Record Dates: First submitted 2021-01-22; First posted 2021-01-26 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-03

CONDITIONS: Myocardial Remodeling After AMI

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acute myocardial infarction patient group (Experimental)
  Interventions: Diagnostic Test: 68Ga-FAPI PET/MRI

INTERVENTIONS:
Diagnostic Test: 68Ga-FAPI PET/MRI — PET and MRI in patients with acute myocardiac infarction are simultaneously analyzed using hybrid PET/MRI device for monitoring myocardial fibrosis and function.

SUMMARY:
Myocardial infarction is the most common cause of high mortality in the modern world. The short-term survival rate of ST-elevated myocardial infarction (STEMI) has been dramatically increased in the past decades thanks to primary coronary intervention and standardization of treatment. However, the long-term prognosis of patients with acute myocardial infarction (AMI) is still poor, especially in the aging population, due to heart failure related to inappropriate myocardial fibrosis and subsequent left ventricular (LV) remodeling. Despite the amelioration of STEMI management, LV remodeling still occurs in approximately 1/3 of all STEMI patients. Therefore, early identification of such patients may help the optimization of therapy and eventually the outcomes.

One characteristic of activated cardiac fibroblasts is the expression of FAP (fibroblast activation protein). A tracer (FAP inhibitor) for positron emission tomography that targets FAP has been used to measure relative FAP density indicative of activated fibroblasts in different cancer entities. However, whether it can reliably assess myocardial fibrosis and predict the poor prognosis caused by LV remodeling is not yet known. Therefore, We aim to observe active myocardial fibrosis process in patients with AMI, and analyze its relationship with the patients'prognosis in a longitudinal study through 68Ga-FAPI PET/MRI.

ELIGIBILITY:
Inclusion Criteria:

* between 18-75 years old
* diagnosed with coronary angiography
* performed percutaneous coronary intervention，with successful myocardial reperfusion

Exclusion Criteria:

* unstable hemodynamics
* MR contraindications (such as pacemaker or nerve stimulator or metal foreign body, high fever, severe renal failure, etc.)
* Claustrophobia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Target-to-background Ratio (TBR) | One week after acute myocardial infarction
  68Ga-FAPI uptake ratio of highly active fibrotic myocardium to heart blood pool on PET images
Metabolic volume (MV) | One week after acute myocardial infarction
  Volume of highly active fibrotic myocardium on PET images
Infarction size (IS) | One week after acute myocardial infarction
  Percentage of late gadolinum enhancement area in the entire myocardium on MRI
Ejection fraction (EF) | One week after acute myocardial infarction
  Left ventricular ejection function evaluated on MRI
Target-to-background Ratio (TBR) | Six months after acute myocardial infarction
  68Ga-FAPI uptake ratio of highly active fibrotic myocardium to heart blood pool on PET images
Metabolic volume (MV) | Six months after acute myocardial infarction
  Volume of highly active fibrotic myocardium on PET images
Infarction size (IS) | Six months after acute myocardial infarction
  Percentage of late gadolinum enhancement area in the entire myocardium on MRI
Ejection fraction (EF) | Six months after acute myocardial infarction
  Left ventricular ejection function evaluated on MRI

SECONDARY OUTCOMES:
NT-pro-BNP | One week after acute myocardial infarction
  Serum marker of chronic heart failure
hsCRP | One week after acute myocardial infarction
  Serum marker of acute myocardial inflammation
NT-pro-BNP | Six months after acute myocardial infarction
  Serum marker of chronic heart failure
hsCRP | Six months after acute myocardial infarction
  Serum marker of acute myocardial inflammation

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ruijin Hospital, Shanghai, China

REFERENCES:
- [Derived] Qiao X, Wang H, Meng H, Xi Y, Feng DD, Li B, Yan X, Zhang M, Huang Q. Multi-modality deep learning-based [68Ga]Ga-DOTA-FAPI-04 PET polar map generation: potential value in detecting reactive fibrosis after myocardial infarction. Eur J Nucl Med Mol Imaging. 2024 Nov;51(13):3944-3959. doi: 10.1007/s00259-024-06850-3. Epub 2024 Jul 26. PMID 39060373